CLINICAL TRIAL: NCT00355407
Title: A Pilot Study of Darbepoetin Alfa (Aranesp) Following Allogeneic Stem Cell Transplantation
Brief Title: Darbepoetin Alfa (Aranesp) Following Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Amgen (Industry); Brigham and Women's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-420
Record Dates: First submitted 2006-07-19; First posted 2006-07-21 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Hematologic Malignancies
Keywords: Aranesp; allogeneic stem cell transplant
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa

SUMMARY:
The purpose of this study is to find out if Darbepoetin alfa is effective in treating low red blood cell levels after allogeneic stem cell transplant. Darbepoetin alfa has been shown to help raise red blood cell levels without blood transfusions.

DETAILED DESCRIPTION:
* Participants will receive Darbepoetin alfa through an injection under the skin, about 28-35 days after their allogeneic stem cell transplant. They will continue to receive the study drug once every three weeks for a maximum of four doses.
* Blood tests will be performed at weeks 3, 6, 9 and 12. The blood tests done at week three will check to make sure the participant has enough iron in their system. If not, they will need to take an iron supplement. Participants will also take a folate supplement to help cell growth and reproduction.

ELIGIBILITY:
Inclusion Criteria:

* Hematologic malignancies undergoing ablative allogeneic stem cell transplantation for any indication
* 18 years of age or older
* Hgb of less than 10 g/dL at the time of initiation therapy

Exclusion Criteria:

* Known hypersensitivity reaction to darbepoetin alfa or any of its components
* Transfusion of packed red blood cells within 3 days of initiation of treatment with darbepoetin alfa
* Any history of grade III or IV GVHD
* Use of any erythropoietic growth factor since transplantation
* Uncontrolled hypertension
* History of seizure
* Baseline creatinine greater than 2
* Dialysis dependence at the time of enrollment
* Hemolytic uremic syndrome
* Active GI bleeding
* Concurrent autoimmune hemolytic anemia
* Concurrent unstable angina
* History of congenital hypercoagulable state or previous venous or arterial thrombosis
* Relapsed disease prior to the initiation of study treatment
* History of renal cell carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31
Dates: Start 2006-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the percentage of patients achieving a target hemoglobin of 11 g/dL or greater by day 100 following allogeneic stem cell transplantation.

SECONDARY OUTCOMES:
Evaluate the percentage of patients achieving a greater than 1 g/dL hemoglobin increase between days 30 and 100 after allogeneic stem cell transplantation
record transfusion requirements between days 30 and 100 in patients undergoing darbepoetin alfa administration following allogeneic stem cell transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jacobsen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States